CLINICAL TRIAL: NCT02847390
Title: Implementation and Evaluation of an Inpatient Diabetes Superuser Education Program
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00071590
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; physician education; nursing education; hyperglycemia; hypoglycemia; inpatient; hospital; glycemic control
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-implementation group: The investigators will develop and deliver a diabetes physician and nursing inpatient diabetes education intervention to our staff over a 6-month time frame from August 2016-January 2017. The investigators will use a before and after study design to assess the impact of the educational intervention on hospital-wide hypoglycemia and hyperglycemia.
  Adult (>18 years), non-obstetrical patients admitted to the medical services where housestaff and hospitalist superusers have been trained, with Type 1 diabetes, Type 2 diabetes, or individuals with hospital-related hyperglycemia who do not carry a prior diabetes diagnosis (4/1/16 to 6/30/16).
- Post-implementation group: Adult (>18 years), non-obstetrical patients admitted to the medical services where housestaff and hospitalist superusers have been trained, with Type 1 diabetes, Type 2 diabetes, or individuals with hospital-related hyperglycemia who do not carry a prior diabetes diagnosis (4/1/17 to 6/30/17).
  Interventions: Other: Education intervention

INTERVENTIONS:
Other: Education intervention — The investigators will develop and deliver a diabetes physician and nursing inpatient diabetes superuser educational curriculum focused on delivering safe, evidence-based diabetes care in the hospital setting. The physician educational curriculum will consist of 10 case-based modules taught to internal medicine residents at two academic hospitals and taught to hospitalists at two academic hospitals and one community hospital. The nursing educational curriculum will consistent of 12 case-based modules taught to unit-based nurses at two academic hospitals and one community hospital. These educational interventions will be delivered over a 6-month time frame from August 2016-April 2017.
  Groups: Post-implementation group

SUMMARY:
The investigators will develop a novel diabetes prescriber superuser educational program focused on inpatient diabetes management for physicians, based on their input. The investigators will then examine the impact of the diabetes prescriber superuser program and an analogous diabetes nurse superuser program that is already developed on glycemic control and other outcomes in hospitalized patients with diabetes.

DETAILED DESCRIPTION:
Both hyperglycemia and hypoglycemia in the hospital are associated with various adverse outcomes, including increased complications, length of stay, cost, and mortality. To address this issue, Johns Hopkins Hospital (JHH) established an Inpatient Glucose Management Program in 2006 to address hypoglycemia and hyperglycemia and to ensure safe, standardized care delivery for hospitalized patients with diabetes. To support nursing education and compliance with JHH glucose management policies, the diabetes nursing "superuser" program was initiated in January 2007 and was critical to implementing the hypoglycemia policy nursing interventions. Following the establishment of hospital-wide glucose management policies and order sets for hypoglycemia and hyperglycemia, the nursing diabetes "superuser" education program, and clinical decision support tools for prescribers, there was a significant and sustained reduction in the incidence of hypoglycemia (~20%) over a 3-year time period. However, the incidence of severe hyperglycemia was not significantly reduced by these interventions, indicating a differential impact of the program on hyperglycemia compared to hypoglycemia. The investigators believe this disparity is due to the hypoglycemia policy being implemented by the nursing staff, whereas the hyperglycemia policy and order set are implemented by prescribers (e.g., housestaff and hospitalists). Given the success of the investigators nursing program's in contributing to sustained reduction in hypoglycemia, the investigators hypothesize that an analogous diabetes prescriber superuser program, targeting physicians, will be an effective educational approach to addressing persistent hyperglycemia. The investigators proposal (1) it seeks to improve diabetes treatment in the hospital, a routine and relevant healthcare setting and (2) it utilizes existing healthcare infrastructure integrated into all hospitals-nursing staff and physicians-making it practical, scalable, and sustainable in other health systems. The investigators have the following specific aims: (1) to develop the diabetes prescriber superuser educational curriculum through Johns Hopkins Health System (JHHS) stakeholder community engagement; (2) to refine and package the JHH diabetes nursing and prescriber superuser educational curricula into an electronic tool kit and disseminate it locally to the 3 JHHS hospitals, based on stakeholder feedback; and (3) to evaluate the impact of implementing the JHH diabetes nursing and prescriber superuser programs at 3 JHHS hospitals on glycemic clinical outcome measures (primary). The investigators will secondarily assess the program's impact on glycemic process and economic measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* non-obstetrical patients admitted to the medical services where housestaff and hospitalist superusers have been trained with Type 1 diabetes or Type 2 diabetes
* individuals with hospital-related hyperglycemia who do not carry a prior diabetes diagnosis

Exclusion Criteria:

* Adults (>18 years) with diabetic ketoacidosis
* hyperosmolar coma
* diabetes with other coma.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years), non-obstetrical patients admitted to the medical services where housestaff and hospitalist superusers have been trained, with Type 1 diabetes, Type 2 diabetes, or individuals with hospital-related hyperglycemia who do not carry a prior diabetes diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 3259 (Actual)
Dates: Start 2015-08; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | Throughout 3 months post intervention
  Percentage and rate of patient-days with at least one hypoglycemic event during admission
Hyperglycemia | Throughout 3 months post intervention
  Percentage of patient-days with patient-day weighted mean blood glucose in hyperglycemia range

CONTACTS AND LOCATIONS:
Overall Officials: Sherita Golden, M.D., M.H.S., Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Golden SH, Hager D, Gould LJ, Mathioudakis N, Pronovost PJ. A Gap Analysis Needs Assessment Tool to Drive a Care Delivery and Research Agenda for Integration of Care and Sharing of Best Practices Across a Health System. Jt Comm J Qual Patient Saf. 2017 Jan;43(1):18-28. doi: 10.1016/j.jcjq.2016.10.004. Epub 2016 Oct 13. PMID 28334581
- [Result] Mathioudakis N, Bashura H, Boyer L, Langan S, Padmanaban BS, Fayzullin S, Sokolinsky S, Hill Golden S. Development, Implementation, and Evaluation of a Physician-Targeted Inpatient Glycemic Management Curriculum. J Med Educ Curric Dev. 2019 Jul 15;6:2382120519861342. doi: 10.1177/2382120519861342. eCollection 2019 Jan-Dec. PMID 31321305